CLINICAL TRIAL: NCT00091026
Title: A Randomized Phase II Study of Bevacizumab (NSC# 704865) and Gemcitabine in Combination With Either Cetuximab (NSC# 714692) or OSI-774 (NSC# 718781) in Patients With Advanced Pancreatic Cancer
Brief Title: Bevacizumab and Gemcitabine Combined With Either Cetuximab or Erlotinib in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02622; NCI-2012-02622 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-6580; UCCRC-13200A; CDR0000383145; 13200A (Other: University of Chicago); 6580 (Other: CTEP); N01CM62204 (NIH); N01CM62203 (NIH); N01CM62201 (NIH); U01CA099118 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2012-12

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Gemcitabine; Bevacizumab; Erlotinib Hydrochloride

ARMS (2):
- Arm I (cetuximab, gemcitabine hydrochloride, bevacizumab) (Experimental): Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, and 22; gemcitabine IV over 30 minutes on days 1, 8, and 15; and bevacizumab IV over 30-90 minutes on days 1 and 15.
  Interventions: Biological: cetuximab; Drug: gemcitabine hydrochloride; Biological: bevacizumab
- Arm II (gemcitabine hydrochloride, bevacizumab, erlotinib) (Experimental): Patients receive gemcitabine and bevacizumab as in arm I. Patients also receive oral erlotinib once daily on days 1-5, 8-12, and 15-26.
  Interventions: Drug: gemcitabine hydrochloride; Biological: bevacizumab; Drug: erlotinib hydrochloride

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
  Arms: Arm I (cetuximab, gemcitabine hydrochloride, bevacizumab)
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
  Arms: Arm II (gemcitabine hydrochloride, bevacizumab, erlotinib)

SUMMARY:
This randomized phase II trial is studying bevacizumab, gemcitabine, and cetuximab to see how well they work compared to bevacizumab, gemcitabine, and erlotinib in treating patients with advanced pancreatic cancer. Monoclonal antibodies, such as cetuximab and bevacizumab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Combining bevacizumab and gemcitabine with either cetuximab or erlotinib may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the objective response rate in patients with advanced adenocarcinoma of the pancreas treated with bevacizumab and gemcitabine with cetuximab vs erlotinib.

II. Compare the toxicity of these regimens in these patients. III. Compare median progression-free and overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center (University of Chicago vs other) and ECOG performance status (0-1 vs 2). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, and 22; gemcitabine IV over 30 minutes on days 1, 8, and 15; and bevacizumab IV over 30-90 minutes on days 1 and 15.

Arm II: Patients receive gemcitabine and bevacizumab as in arm I. Patients also receive oral erlotinib once daily on days 1-5, 8-12, and 15-26.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 54-126 patients (27-63 per treatment arm) will be accrued for this study within 16 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Advanced disease

    * Patients with locally advanced disease must have disease that extends outside the boundaries of a standard radiation port
* Not amenable to curative surgery or radiotherapy
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
  * Pleural effusions and ascites are not considered measurable lesions
* No CNS disease, including primary brain tumors or brain metastasis
* No tumor invasion into the duodenum
* Performance status - ECOG 0-2
* More than 3 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,000/mm^3
* No history of bleeding diatheses
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT and SGPT ≤ 2.5 times ULN (5 times ULN if liver metastases are present)
* INR ≤ 1.5 (≤ 3 for patients on warfarin)
* No esophageal varices
* Creatinine ≤ 1.5 mg/dL
* Creatinine clearance ≥ 60 mL/min
* Urine protein < 1+
* 24-hour urine protein < 500 mg
* No history of a recent cerebrovascular accident
* No clinically significant cardiovascular disease
* No uncontrolled hypertension
* No New York Heart Association class II-IV congestive heart failure
* No serious cardiac arrhythmia requiring medication
* No peripheral vascular disease ≥ grade II
* None of the following arterial thromboembolic events within the past 6 months:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina
  * Myocardial infarction
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study participation
* HIV negative
* No significant traumatic injury within the past 28 days
* No gastrointestinal tract disease resulting in an inability to take oral medication
* No allergic reactions to compounds similar to bevacizumab, cetuximab, or erlotinib (e.g., Chinese hamster ovary cell products or recombinant humanized antibodies)
* No serious or non-healing wound, ulcer, or bone fracture
* No active infection requiring antibiotics
* No other active malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No prior bevacizumab or cetuximab
* No other prior vascular endothelial growth factor inhibitors
* No prior gemcitabine
* No prior cytotoxic chemotherapy for metastatic disease
* At least 4 weeks since prior adjuvant chemotherapy (6 weeks for mitomycin or nitrosoureas)
* At least 4 weeks since prior radiotherapy

  * Must have a site of measurable disease outside the radiation port
* No prior surgical procedure affecting absorption
* More than 28 days since prior major surgical procedure or open biopsy
* More than 7 days since prior core biopsy
* No concurrent major surgical procedures
* No prior erlotinib
* No other prior epidermal growth factor receptor inhibitors
* At least 30 days since prior investigational drugs
* More than 1 month since prior thrombolytic agents
* Concurrent warfarin or low molecular weight heparin allowed provided the following criteria are met:

  * Currently therapeutic on a stable dose
  * INR target range ≤ 3
  * Patients undergo weekly INR testing
  * No evidence of active bleeding or pathological condition that carries high risk of bleeding (e.g., tumor invading adjacent organs or esophageal varices)
* No concurrent chronic daily therapy with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory medications known to inhibit platelet function
* No other concurrent antiplatelet medications
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapies or agents
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2004-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at sixteen sites between September 2004 and February 2007.
Period: Overall Study
Arm/Group | Arm I (Cetuximab, Gemcitabine Hydrochloride, Bevacizumab) | Arm II (Gemcitabine Hydrochloride, Bevacizumab, Erlotinib)
Started | 72 | 71
Completed | 71 | 68
Not Completed | 1 | 3
Not completed — Patient deemed non eligible-never receiv | 1 | 0
Not completed — Patient withdrew and never received trea | 0 | 2
Not completed — Unknown-never received treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: Four patients who never received treatment are excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Cetuximab, Gemcitabine Hydrochloride, Bevacizumab) | Arm II (Gemcitabine Hydrochloride, Bevacizumab, Erlotinib) | Total
Number analyzed (Participants) | 71 | 68 | 139
Age, Continuous [Median (Full Range); unit: years] | 63 [36 to 83] | 63 [39 to 86] | 63 [36 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 19 | 56
  Male | 34 | 49 | 83
ECOG Performance Status [Number; unit: Participants] — ECOG Performance Status
  The scale ranges from 0-5:
  0 Fully active, without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities.
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
  Participants
    0 | 26 | 32 | 58
    1 | 40 | 32 | 72
    2 | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Complete or Partial Response) Evaluated Using the Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: Up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Cetuximab, Gemcitabine Hydrochloride, Bevacizumab) | Arm II (Gemcitabine Hydrochloride, Bevacizumab, Erlotinib)
Number analyzed (Participants) | 71 | 68
percentage of participants | 21 [12 to 32] | 21 [12 to 32]
Statistical Analysis 1: Comparison: Arm I (Cetuximab, Gemcitabine Hydrochloride, Bevacizumab) vs Arm II (Gemcitabine Hydrochloride, Bevacizumab, Erlotinib); Test type: Superiority or Other; p = 0.22, Chi-squared; Risk Difference (RD) = 0, 95% CI 2-sided [-13 to 14]

2. Secondary Outcome: Progression-free Survival
Description: Median progression-free survival time (time from randomization to disease progression or death from any cause). Analyzed using the Kaplan-Meier (1958) estimator and their associated 95% confidence intervals determined using the method described in Brookmeyer and Crowley.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Cetuximab, Gemcitabine Hydrochloride, Bevacizumab) | Arm II (Gemcitabine Hydrochloride, Bevacizumab, Erlotinib)
Number analyzed (Participants) | 71 | 68
months | 5.0 [3.7 to 5.5] | 5.1 [3.2 to 5.9]
Statistical Analysis 1: Comparison: Arm I (Cetuximab, Gemcitabine Hydrochloride, Bevacizumab) vs Arm II (Gemcitabine Hydrochloride, Bevacizumab, Erlotinib); Test type: Superiority or Other; p = 0.95, Log Rank

3. Secondary Outcome: Overall Survival
Description: Time from randomization until death from any cause. Analyzed using the Kaplan-Meier (1958) estimator and their associated 5% confidence intervals determined using the method described in Brookmeyer and Crowley.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Cetuximab, Gemcitabine Hydrochloride, Bevacizumab) | Arm II (Gemcitabine Hydrochloride, Bevacizumab, Erlotinib)
Number analyzed (Participants) | 71 | 68
Months | 7.9 [5.5 to 9.5] | 7.1 [5.4 to 9.1]
Statistical Analysis 1: Comparison: Arm I (Cetuximab, Gemcitabine Hydrochloride, Bevacizumab) vs Arm II (Gemcitabine Hydrochloride, Bevacizumab, Erlotinib); Test type: Superiority or Other; p = 0.86, Log Rank

ADVERSE EVENTS:
Arm/Group | Arm I (Cetuximab, Gemcitabine Hydrochloride, Bevacizumab) | Arm II (Gemcitabine Hydrochloride, Bevacizumab, Erlotinib)
Serious Adverse Events (participants affected / at risk) | 21/71 | 17/68
Other Adverse Events (participants affected / at risk) | 57/71 | 44/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Cetuximab, Gemcitabine Hydrochloride, Bevacizumab) (N=71) | Arm II (Gemcitabine Hydrochloride, Bevacizumab, Erlotinib) (N=68)
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Abdominal cramping (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 | 0
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Bladder infection (Infections and infestations) | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1
CVA (Vascular disorders) | 3 | 0
Cholecystitis NOS (Hepatobiliary disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Fatigue (General disorders) | 1 | 2
GI bleeding (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Hematoma (Vascular disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 2 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 2 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Left ventricular failure (Cardiac disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 1
Nausea/vomiting (Gastrointestinal disorders) | 1 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Syncope/vasovagal (Nervous system disorders) | 0 | 1
Thrombosis/embolism (Vascular disorders) | 4 | 2
Thrombotic microangiopathy (Vascular disorders) | 0 | 1
Vascular access complication (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Cetuximab, Gemcitabine Hydrochloride, Bevacizumab) (N=71) | Arm II (Gemcitabine Hydrochloride, Bevacizumab, Erlotinib) (N=68)
Anorexia (Metabolism and nutrition disorders) | 5 | 2 — Worst grade 3 or higher and at least possibly related to treatment
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 3 | 8 — Worst grade 3 or higher and at least possibly related to treatment
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 0 | 4 — Worst grade 3 or higher and at least possibly related to treatment
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 3 | 6 — Worst grade 3 or higher and at least possibly related to treatment
Dehydration (Metabolism and nutrition disorders) | 2 | 5 — Worst grade 3 or higher and at least possibly related to treatment
Diarrhea (Gastrointestinal disorders) | 2 | 4 — Worst grade 3 or higher and at least possibly related to treatment
Fatigue (General disorders) | 11 | 9 — Worst grade 3 or higher and at least possibly related to treatment
Hemoglobin (Blood and lymphatic system disorders) | 2 | 6 — Worst grade 3 or higher and at least possibly related to treatment
Nausea/vomiting (Gastrointestinal disorders) | 5 | 6 — Worst grade 3 or higher and at least possibly related to treatment
Neutropenia (Investigations) | 18 | 21 — Worst grade 3 or higher and at least possibly related to treatment
Platelet count decreased (Investigations) | 10 | 15 — Worst grade 3 or higher and at least possibly related to treatment
Proteinuria (Renal and urinary disorders) | 1 | 4 — Worst grade 3 or higher and at least possibly related to treatment
Rash/dermatitis (Skin and subcutaneous tissue disorders) | 8 | 3 — Worst grade 3 or higher and at least possibly related to treatment
Thrombosis/embolism (Vascular disorders) | 5 | 2 — Worst grade 3 or higher and at least possibly related to treatment
White blood cell count (Investigations) | 9 | 9 — Worst grade 3 or higher and at least possibly related to treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less